CLINICAL TRIAL: NCT07004153
Title: A Multicenter, Open Label, Randomized, Comparative Confirmatory Study to Evaluate the Efficacy and Safety of Electric Smart Insulin Pen (DIA:CONN P8) Including Setup Wizard, Advanced Insulin Injection Coaching and Bolus Calculator With Analysis Function Based on Continuous Glucose Monitoring Data in Patients With Type 1 or Type 2 Diabetes Mellitus Under Multiple Dose Insulin Therapy
Brief Title: A Study of DIA:CONN P8 Smart Insulin Pen With CGM-Based Coaching in Patients With Type 1 or Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G2e Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P8_S201
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Group (Experimental): Basal and bolus insulin injection using an electric smart insulin pen (DIA:CONN P8); equipped with a Setup-wizard, CGM-based Advanced insulin injection Coaching and a Bolus calculator
  - Providing education on Carb Counting(carbohydrate measurement) and Methods for adjusting insulin bolus calculator
  Interventions: Device: Smart Coaching Insulin Pen
- Control group (No Intervention): Basal and bolus insulin injection using only the injection and recording functions of DIA:CONN P8
  - Subjects manually enter and inject their insulin doses without using the bolus calculator or coaching functions

INTERVENTIONS:
Device: Smart Coaching Insulin Pen — Subjects randomized to the intervention group will use the DIA:CONN P8 smart insulin pen with full functionality, including Setup Wizard, CGM-based insulin injection coaching, and a bolus calculator. During the 12-week application period, including the baseline visit, participants will visit the hospital up to 5 times. At the start of the period, initial basal and bolus doses will be determined using the Setup Wizard and reviewed by investigators. Throughout the study, subjects will receive real-time insulin dose recommendations and coaching via the DIA:CONN app based on CGM data, carbohydrate input, and insulin dosing history.
  Arms: Investigational Group

SUMMARY:
A Study of DIA:CONN P8 Smart Insulin Pen With CGM-Based Coaching in Patients With Type 1 or Type 2 Diabetes

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of the DIA:CONN P8, an electric smart insulin pen equipped with a Setup Wizard, CGM-based insulin injection coaching, and a bolus calculator. The device is designed to support patients with type 1 or type 2 diabetes who are on multiple daily insulin injections (MDI). The study compares the outcomes of patients using these advanced features to those using only the injection and recording functions of the device.

The rationale stems from previous research showing that structured education in combination with CGM improves glycemic control in patients with diabetes. The DIA:CONN P8 aims to replicate the benefits of such structured education through app-based coaching and algorithm-driven recommendations, potentially reducing the burden of complex insulin dose calculations in routine care.

Participants will undergo a run-in period using DIA:CONN P8 with injection-only functionality to assess compliance. Eligible subjects will then be randomized into either the investigational group (using all device functions) or the control group (injection and recording only). Over 12 weeks, the primary endpoint is the change in HbA1c. Secondary outcomes include CGM-based metrics such as Time in Range (TIR), Time Below Range (TBR), and insulin dosing behavior.

The study is designed as a multicenter, open-label, randomized, comparative confirmatory trial conducted at six sites. A total of 152 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 19 and 75 years old.
2. Diagnosis of type 1 or type 2 diabetes for at least 1 year prior to screening
3. Continuous use of MDI therapy for at least 3 months prior to screening, defined as one of the following regimens:

   * Long-acting insulin plus rapid-/short-acting insulin
   * Mixed insulin (e.g., insulin aspart/insulin degludec) plus rapid-/short-acting insulin
   * Mixed insulin ≥3 times per day
4. HbA1c of 7.5% to 12.0% at screening.

Exclusion Criteria:

1. Diabetes mellitus secondary to pancreatic resection.
2. Use of corticosteroids exceeding a prednisolone-equivalent dose of 5 mg/day within 3 months prior to screening (Subjects on a stable dose for ≥3 months prior to screening may be eligible).
3. eGFR <15 mL/min at screening or those receiving dialysis
4. Pregnant or lactating women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c(%) at 12 weeks compared to baseline | from baseline to the 12-week time point
  Descriptive statistics (sample size, mean, standard deviation, median, minimum, and maximum) are provided for the change in HbA1c (%) from baseline to the 12-week time point, stratified by group.

CONTACTS AND LOCATIONS:
Overall Officials: TAEMIN LEE, Study Director — G2e Co., Ltd
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JY, Kim NH, Kwak SH, Jung CH, Kang ES, Moon JS, Moon SJ, Kwon SY, Yoo JH, Kim Y, Lee TM, Yang CI, Kim JH, Jin SM. Efficacy and Safety of Stage 5 Connected Insulin Pens in Type 1 or Type 2 Diabetes: Randomized Controlled Trial Protocol. Endocrinol Metab (Seoul). 2025 Dec 12. doi: 10.3803/EnM.2025.2579. Online ahead of print. PMID 41391451